CLINICAL TRIAL: NCT02041013
Title: The Talking Card for Asthma: A Recordable Audio Discharge Instruction Device to Improve Asthma Control
Brief Title: Talking Card for Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: University of South Florida (Other)
Responsible Party: Principal Investigator, John D Cowden, Associate Professor of Pediatrics, Children's Mercy Hospital Kansas City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 0909209E
Record Dates: First submitted 2014-01-17; First posted 2014-01-20 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Asthma
Keywords: Asthma; Health Literacy
MeSH Terms: conditions — Asthma

ARMS (2):
- No Talking Card (No Intervention): Usual care of asthma by study clinician, including evaluation of asthma using C-ACT and clinical history, treatment using asthma action planning
- Taking Card (Experimental): Usual care, as in comparison group, plus recordable Talking Card at each visit
  Interventions: Other: Taking Card

INTERVENTIONS:
Other: Taking Card — Recordable greeting card-style discharge instruction card
  Arms: Taking Card

SUMMARY:
The research goal is to explore the use and effects of a custom-recordable audio discharge instruction card (Talking Card) in the pediatric health care setting. This study will address a primary, experimental research question: can pediatric asthma control be improved through the distribution of a custom-recorded audio asthma instruction card to parents at the health provider's office? Secondary, descriptive objectives will be to evaluate feasibility of Talking Card delivery and to collect and summarize parental reactions to the design and use of the audio discharge instruction card.

The specific aims of this study are:

1. To compare the change in mean Childhood Asthma Control Test (C-ACT) scores for children aged 4 through 11 years with uncontrolled asthma receiving a custom-recorded asthma instruction card to the change in mean C-ACT scores for those receiving usual care.
2. To measure the use and impressions of a custom-recordable audio asthma discharge instruction card among primary caregivers of children with uncontrolled asthma through quantitative and qualitative survey questions.

The investigators hypothesize that:

1) Asthma control in children 4 through 11 years of age with uncontrolled asthma, as measured by the C-ACT, will improve to a greater extent among those receiving a custom-recordable audio discharge instruction card than among those receiving usual care.

ELIGIBILITY:
Inclusion Criteria:

* Child age 4 through 11 years old
* English-speaking primary caregiver
* Enrollment in Medicaid insurance company within 12 months of study recruitment (original Kansas City site criterion, removed on revision)
* Diagnosis of asthma (ICD-9 code 493.0) within 12 months of study recruitment
* Visit to study site clinic for asthma within 12 months of study recruitment

Exclusion Criteria:

* History of premature birth less than 33 weeks gestation or requirement of a significant level of respiratory care including mechanical ventilation as a neonate
* Any major chronic illness including but not limited to non-skin cancer, cystic fibrosis, bronchiectasis, sickle cell anemia, endocrine disease, congenital heart disease, congestive heart failure, stroke, severe hypertension, insulin-dependent diabetes mellitus, renal failure, liver disorders, immunodeficiency states, significant neuro-developmental delay or behavioral disorders (excluding mild attention deficit hyperactivity disorder), or other conditions that would interfere with participation in the study
* Visit to any primary care provider giving asthma action plan advice during the previous month
* Anticipated departure from study area before study period ends (3-month follow-up)

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2009-11; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Asthma Control (C-ACT) | 3 months
  Childhood Asthma Control Test (C-ACT) score, measured repeatedly across 3 visits

SECONDARY OUTCOMES:
Parental Card Use and Satisfaction | 3 months
  Survey of parental card use and satisfaction with card performance, measured repeatedly across 3 visits

CONTACTS AND LOCATIONS:
Overall Officials: John D Cowden, MD,MPH, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (2):
- United States (2):
  - University of South Florida, Tampa, Florida
  - Children's Mercy Hospital, Kansas City, Missouri